CLINICAL TRIAL: NCT01478282
Title: Evaluation of the Potential Action of Coagulation Factors Concentrates in the Reversal of the Antithrombotic Action of New Oral Anticoagulants: Studies ex Vivo in Blood Samples From Healthy Volunteers
Brief Title: Reversal of the Antithrombotic Action of New Oral Anticoagulants
Acronym: REVANT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gines Escolar (Other)
Collaborators: Ministry of Health, Spain (Other Government)
Responsible Party: Sponsor-Investigator, Gines Escolar, head of department Hemotherapy-Hemostasis, Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Single
Other Study IDs: FCRB; 2010-022985-29 (EudraCT Number)
Record Dates: First submitted 2011-11-08; First posted 2011-11-23 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Thrombosis; Anticoagulant-induced Bleeding; Anticoagulant Overdosage; Hemorrhage
Keywords: dabigatran; rivaroxaban; oral anticoagulants; coagulation; bleeding; plasma concentrates
MeSH Terms: conditions — Thrombosis; Hemorrhage | interventions — Rivaroxaban; Dabigatran

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rivaroxaban (Active Comparator): Healthy donors subjected to 20mg/day for 5 days
  Interventions: Drug: Rivaroxaban
- Dabigatran (Active Comparator): Healthy volunteers subjected to 150 mg/12hours for 5 days
  Interventions: Drug: Dabigatran

INTERVENTIONS:
Drug: Rivaroxaban — 20 mg/day, oral administration maintained for 5 days
  Other Names: Xarelto is the brand name for rivaroxaban
  Arms: Rivaroxaban
Drug: Dabigatran — 150 mg/12 hours, administered orally, treatment maintained for 5 days
  Other Names: Pradaxa is the brand name for dabigatran
  Arms: Dabigatran

SUMMARY:
The main goal of this study is to improve safety and efficiency of clinical practice with the new generation of oral anticoagulants.

1. To determine the effect of new oral anticoagulants (dabigatran and rivaroxaban) on platelets and coagulation mechanisms under flow conditions.
2. To evaluate the ability of the concentrates containing coagulation factors (PCCs and FVIIa) to reverse the effects induced by the new anticoagulants.

These studies will be carried out ex vivo in blood samples obtained from healthy volunteers undergoing oral anticoagulant therapy at doses of proven efficacy and safety used in previous clinical trials.

DETAILED DESCRIPTION:
There is a lack of information on antidotes that could reverse the effects of new oral anticoagulants in patients that require a rapid restoration of their impaired hemostatic mechanisms. The present study seeks to improve the security and efficacy of the clinical practice with the new generation of oral anticoagulants.

OBJECTIVES:

1. To assess the action of new oral anticoagulants (dabigatran y rivaroxaban) on hemostasis with specific interest on possible interference with platelet interactions and coagulation mechanisms under flow conditions;
2. To evaluate comparatively the effects of coagulation factor concentrates of established efficacy (prothrombin complexes and rFVIIa) to reverse the alterations of hemostasis parameters induced by the new anticoagulants.

METHODOLOGY:

Studies will be performed ex vivo using blood samples from healthy individuals subjected to treatments with the new anticoagulants at doses of proven efficacy and safety (150mg/12 h for dabigatran and 20 mg/day for rivaroxaban). Blood samples from the participants will be spiked "in vitro" with know concentrations of the coagulation factors. Modifications in:

* morphometric parameters (platelet deposition and fibrin formation) in perfusion studies under flow conditions; and
* analytical tests evaluating changes in coagulation mechanisms (thrombin generation, ecarine and prothrombin times) will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers ages from 21 to 60 years
* Approval informed consent

Exclusion Criteria:

* History of hepatic or kidney disease
* Previous history of hemorrhagic or thrombotic disease
* Pregnancy or breast feeding
* Concomitant use of drugs affecting hemostasis
* Use of medications of herbal treatments that could interfere with the pharmacokinetics or pharmacodynamics of the study drug (according to manufacturers label)
* Practice of risky sports (during the study period)
* Blood donation in the previous 3 months

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Modifications in hemostasis parameters. | 5 days
  We will evaluate: a) the surface covered by platelets and fibrin on the subendothelium of vascular segments. Platelet interaction will be expressed as percentage of covered surface by platelets (%CS) and classified as contact, adhesion and aggregates depending of the size of interactions. Fibrin formation will be also evaluated as percentage of surface covered by fibrin (%F) and as the mean area of fibrin formed; and b) thrombin generation as lag time and maximum thrombin peak generation using a commercially available test (Technothrombin TGA, Technoclone GMBH).
Changes observed after in vitro addition of coagulation factor concentrates | 5 days
  We will re-evaluate: a) the surface covered by platelets and fibrin on the subendothelium of vascular segments. Platelet interaction will be expressed as percentage of covered surface by platelets (%CS) and classified as contact, adhesion and aggregates depending of the size of interactions. Fibrin formation will be also evaluated as percentage of surface covered by fibrin (%F) and as the mean area of fibrin formed; and b) thrombin generation as lag time and maximum thrombin peak generation using a commercially available test (Technothrombin TGA, Technoclone GMBH).

SECONDARY OUTCOMES:
Measure other indirect biomarkers of the activation of the coagulation mechanisms. | 5 days
  Prothrombin time, ecarin clotting time, and F1+2 fragments will be determined in frozen plasma samples.

CONTACTS AND LOCATIONS:
Overall Officials: Gines Escolar, M.D., Ph.D., Principal Investigator — Fundacio Clinic per a la Reçerca Biomedica (FCRB)
Locations (1):
- Hospital Clinic, Fundació Clinic (FCRB), Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Arellano-Rodrigo E, Lopez-Vilchez I, Galan AM, Molina P, Reverter JC, Carne X, Villalta J, Tassies D, Lozano M, Diaz-Ricart M, Escolar G. Coagulation Factor Concentrates Fail to Restore Alterations in Fibrin Formation Caused by Rivaroxaban or Dabigatran in Studies With Flowing Blood From Treated Healthy Volunteers. Transfus Med Rev. 2015 Oct;29(4):242-9. doi: 10.1016/j.tmrv.2015.08.001. Epub 2015 Aug 8. PMID 26364029